CLINICAL TRIAL: NCT03967262
Title: Secondary Prevention and Recidivism Reduction in Trauma Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Salvador Navarro-Soto, Head of General and Digestive Surgery Department, Corporacion Parc Tauli
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CSPT-CG-PPT2
Record Dates: First submitted 2019-05-26; First posted 2019-05-30 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Trauma; Alcohol Use, Unspecified; Drug Use
MeSH Terms: conditions — Wounds and Injuries; Alcohol Drinking

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Behavioral: Brief Motivational Intervention
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Brief Motivational Intervention — The objective of motivational intervention is to make the patient aware of the relationship between the consumption of alcohol and other drugs and the accident, and induce them to carry out a change in habits.
  Arms: Intervention

SUMMARY:
The consumption of alcohol and other drugs is one of the main risk factors for traumatism. In addition, patients who have suffered an accident in relation to the consumption of these substances present a high risk of recidivism. In the case of alcohol, its relationship with traumatisms has been known for many years now and is still one of the main risk factors.

Secondary prevention is an important area of action and improvement in the treatment of this type of patient by considering actions, such as a brief motivational intervention, in order to avoid recidivism. The objective of motivational intervention is to make the patient aware of the relationship between the consumption of these substances and the accident, and induce them to carry out a change in habits.

The objective of the present investigation project is to determine the efficacy of secondary prevention in reducing recurrence of traumatisms. In order to this, a multicenter randomised controlled trial has been designed in which the intervention group with patients admitted for sever traumatism with positive screening for alcohol or other drugs, will be submitted to a brief motivational intervention. The main outcome will be trauma recurrence within a three year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Sever trauma patients defined as the need of assistance in a critical unit.
* Positive screening for alcohol o other drugs (cannabis, cocaine, methamphetamine).

Exclusion Criteria:

* Patients in treatment for abuse of alcohol and other drugs.
* Death during hospitalization.
* Non Catalonia residents.
* Not Spanish or Catalan spoken.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence of traumatisms | Follow-up of 3 years
  Any medical assistance related to a traumatism

SECONDARY OUTCOMES:
Alcohol prevalence | Trough study completion, an average of 2 years
  Alcohol prevalence among trauma patients
Other drugs prevalence (cannabis, cocaine, methamphetamine) | Trough study completion, an average of 2 years
  Other drugs prevalence among trauma patients
Time to a recurrence | Trough study completion, an average of 2 years
  Time since discharge until the first new trauma or withdrawal from follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Salvador Navarro-Soto, PhD, Principal Investigator — Corporacion Sanitaria Parc Tauli; Salvador Navarro-Soto, PhD, Study Director — Corporacion Sanitaria Parc Tauli
Locations (1):
- Corporacion Sanitaria Parc Taulí, Sabadell, Barcelona, Spain